CLINICAL TRIAL: NCT04932993
Title: Writing Down Goals
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Deemed not feasible.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, David Ring, MD, PhD Associate Dean for Comprehensive Care, Professor of Surgery and Psychiatry, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-07-0089
Record Dates: First submitted 2021-06-08; First posted 2021-06-21 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Musculoskeletal Diseases
Keywords: decisional conflict; Orthopedics
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: All new, adult (18+ years old) patients seeing an orthopedic surgeon for a consultation will be invited to participate in this study. Patients randomly will be assigned to: write down goals their goals for their medical care (intervention) or not (usual visit control group). The research assistant will ask the patient to fill out a survey entailing demographics, JSPPE, the communication effectiveness score, the PAM score and a satisfaction scale at the end of the visit. A research assistant will record the diagnosis,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Will not write down goals their goals for their medical care (usual care).
- Writing down goals (Experimental): Will write down goals their goals for their medical care.
  Interventions: Behavioral: Writing down goals

INTERVENTIONS:
Behavioral: Writing down goals — Patient will write their health goals down before the visit.
  Arms: Writing down goals

SUMMARY:
The women's health IPU at UT Health Austin is happy with having patients write down their goals at their first visit and then tracking those. It would be interesting to study people seeking musculoskeletal specialty care to determine whether asking patients what result of their care would be rated a success helps direct the clinician-patient interaction in a more fruitful direction compared to the usual clinical interaction.

DETAILED DESCRIPTION:
People's stated preferences are often inconsistent with what matters most to them (their values). And they are often based on misconceptions, distress, and less effective cognitive coping strategies. For instance, a person might say "My goal is to have no pain" when that is not possible. Or they might say "My goal is to get the shot that fixes this" when there is no such shot. It may go without saying that people want: "To be able to live a normal lifestyle" and "To be able to accomplish most of their goals." In other words, people want to be able to be themselves. They are seeking care because they are not able to be themselves or they are concerned that they may not be able to be themselves. The word health comes from an old German word meaning "whole."

One part of good health is correcting or alleviating pathophysiology (e.g. reading glasses). Another part of good health is evolving one's inner narrative (e.g. "I'm older now and need glasses to read").

The women's health IPU at UT Health Austin is happy with having patients write down their goals at their first visit and then tracking those. It would be interesting to study people seeking musculoskeletal specialty care to determine whether asking patients what result of their care would be rated a success helps direct the clinician-patient interaction in a more fruitful direction compared to the usual clinical interaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+)
* Orthopedic visit

Exclusion Criteria:

* Patients who are illiterate.
* Patients who do not speak English.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Decision conflict questionnaire | Baseline
  Questionnaire assessing decision conflict

SECONDARY OUTCOMES:
Decision regret questionnaire | Baseline
  Questionnaire assessing the degree of regret of decision
Jefferson Scale of Patient's Perceptions of Physician Empathy | Baseline
  Patient perceived of physician empathy as measured by the JSPPE
Patient Activation Measure-13 | Baseline
  Patient activation as measured by PAM-13
Guttman Satisfaction scale | Baseline
  Questionnaire measuring to what degree patients are satisfied with the care they received.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Professor of Surgery, Dell Medical School at The University of Texas at Austin

IPD SHARING:
Plan to Share IPD: No